CLINICAL TRIAL: NCT02965573
Title: A Randomized, Double-blind, Placebo-Controlled Phase II Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of ARGX-113 in Patients With Myasthenia Gravis Who Have Generalized Muscle Weakness
Brief Title: A Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of ARGX-113 in Patients With Myasthenia Gravis Who Have Generalized Muscle Weakness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: argenx (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARGX-113-1602; 2016-002938-73 (EudraCT Number)
Record Dates: First submitted 2016-10-20; First posted 2016-11-17 (Estimated); Results first posted 2021-01-08 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — efgartigimod alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARGX-113 (Active Comparator): During the Treatment period, eligible patients will be randomized at a 1:1 ratio to receive ARGX-113
  Interventions: Biological: ARGX-113
- Placebo (Placebo Comparator): During the Treatment period, eligible patients will be randomized at a 1:1 ratio to receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: ARGX-113
  Arms: ARGX-113
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicenter Phase II study to evaluate the safety, efficacy, and pharmacokinetics of ARGX-113 for the treatment of autoimmune Myasthenia Gravis (MG) with generalized muscle weakness.

DETAILED DESCRIPTION:
Myasthenia Gravis (MG) is an autoimmune disorder characterized in most cases by T cell and antibody responses to neuromuscular junction proteins such as skeletal muscle nicotinic acetylcholine receptor (AChR). Antibodies against epitopes of the AChR of the neuromuscular junction cause failure of neuromuscular transmission, resulting in the characteristic fatigue and weakness associated with this severe disorder.

The study will evaluate an innovative candidate in MG.

ELIGIBILITY:
Inclusion Criteria:

1. Have the ability to understand the requirements of the study, provide written informed consent (including consent for the use and disclosure of research-related health information), and comply with the study protocol procedures (including required study visits).
2. Male or female patients aged ≥18 years.
3. Diagnosis of autoimmune MG with generalized muscle weakness meeting the clinical criteria for diagnosis of MG as defined by the Myasthenia Gravis Foundation of America (MGFA) Clinical Classification Class II, III, or IVa, and likely not in need of a respirator for the duration of the study as judged by the Investigator.

   The confirmation of the diagnosis should be documented and supported by:
   * Positive serologic test for anti-AChR antibodies before Screening and
   * at least 1 of the following 3 tests: (i) History of abnormal neuromuscular transmission test demonstrated by single-fiber electromyography or repetitive nerve stimulation or (ii) History of positive edrophonium chloride test, or (iii) Patient has demonstrated improvement in MG signs on oral cholinesterase inhibitors as assessed by the treating physician.
4. A total score of ≥ 5 on the MG ADL at Screening and Baseline with more than 50% of this score attributed to non ocular items.
5. Patients are required to be on a stable dose of their MG treatment prior to randomization. For patients receiving AZA, other NSIDs, steroids, and/or cholinesterase inhibitors as concomitant medications the following conditions will apply:

   * AZA: treatment initiated at least 12 months ago and no dose changes in the last 6 months before screening.
   * Other NSIDs (e.g., methotrexate, cyclosporine, tacrolimus, mycophenolate mofetil, and cyclophosphamide) treatment initiated at least 6 months ago and no dose changes in the last 3 months before Screening.
   * Steroids treatment initiated at least 3 months prior to and no dose changes in the last month before Screening.
   * Cholinesterase inhibitors: to be on a stable dose for >2 weeks before Screening.

   Note: cholinesterase inhibitors must be held for at least 12 hours consistent with the revised manual for the QMG test as recommended by the Myasthenia Gravis Foundation of America Inc (MGFA), before the MGQoL15r, MG-ADL, QMG, and MGC assessments.
6. Females of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Visit 1 prior to administration of IMP. Female of childbearing potential are defined as all female participants unless they are postmenopausal (defined by continuous amenorrhea) for at least 2 years with a Follicle stimulating hormone (FSH) > 40 IU/L or are surgically sterile (i.e., who had a hysterectomy, bilateral oophorectomy, or have current documented tubal ligation or any other permanent female sterilization procedure). Determination of FSH levels can be used to confirm postmenopausal status in amenorrheic patients not on hormonal replacement therapy if the test result is within the postmenopausal range per the central laboratory.
7. Female participants of childbearing potential must agree to use a highly effective method of contraception (i.e., pregnancy rate of less than 1% per year) during the study and for 90 days after the discontinuation of the IMP. Adequate contraceptive methods include combined hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine devices (IUDs), intrauterine hormone-releasing system (IUS), true sexual abstinence (when this is in line with the preferred and usual lifestyle of the participant), bilateral tubal occlusion, or a female participant who is not of childbearing potential. Female participants and female partners of male study participants using a hormonal contraceptive must also use a barrier method (i.e., condom or occlusive cap [diaphragm or cervical/vault caps]) and should have been stable on their hormonal contraceptive treatment for at least 4 weeks before Screening.
8. Sterilized male patients who have had vasectomy with documented aspermia post procedure can be included. In addition, male patients must be advised not to donate sperm during this period from signing of Informed Consent Form (ICF), throughout the duration of the study, and for 90 days after the last administration of IMP. Non-sterilized male patients who are sexually active with a female partner of childbearing potential must use effective method of double barrier contraception (e.g., condom with spermicidal cream or jelly, 1 hormonal plus 1 barrier method or 2 simultaneous barrier methods). Male patients practicing true sexual abstinence (when this is in line with the preferred and usual lifestyle of the participant) can be included.

Exclusion Criteria:

1. Females who are pregnant or lactating.
2. MGFA Class I, IVb, and V.
3. Have an active infection, a recent serious infection (i.e., requiring injectable antimicrobial therapy or hospitalization) within the 8 weeks prior to Screening; or history of or known infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), or Mycobacterium tuberculosis. Patients must have negative test results for HBV surface antigen, HBV core antibody, HCV antibody, HIV 1 and 2 antibodies, and a negative QuantiFERON®-TB Gold test at Screening. Patients with an indeterminate QuantiFERON®-TB Gold test result will be allowed one retest; if not negative on retesting, the patient will be excluded.
4. At Screening, have clinically significant laboratory abnormalities or as below:

   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) > 2 x upper limit of normal (ULN).
   * Total serum bilirubin of > 1.5 x ULN (except for Grade 1 hyperbilirubinemia solely due to a medical diagnosis of Gilbert's syndrome).
   * Serum creatinine > 1.5 mg/dL and creatinine clearance < 50 ml/min (using the Chronic Kidney Disease Epidemiology [CKD-EPI]-Creatinine formula).
   * Clinically Significant proteinuria (i.e., > 3 x ULN).
   * Hemoglobin ≤ 9 g/L.
   * Thyroid stimulating hormone or thyroglobulin outside of the central laboratory normal range.
   * International normalized ratio (INR) or activated partial thromboplastin time (aPTT) > 1.2 x ULN.
   * Total immunoglobulin G level < 6 g/L.
5. Body Mass Index (BMI) at Screening ≥ 35 kg/m2.
6. Use of rituximab, belimumab, eculizumab or any monoclonal antibody for immunomodulation within 6 months prior to first dosing. Patients with prior exposure to rituximab must have CD19 counts within the normal range per the central laboratory at Screening.
7. Use of any biological therapy or investigational drug within 3 months or 5 half-lives of the drug (whichever is longer) before Screening.
8. Immunoglobulins given by IV (IVIg), or intramuscular route, or plasmapheresis/plasma exchange (PE) within 4 weeks before Screening.
9. Have known autoimmune disease other than MG that would interfere with the course and conduct of the study (such as uncontrolled thyroid disease or severe RA).
10. Have received vaccinations within 4 weeks before Screening or have any vaccinations planned during the study.
11. Have a history of malignancy, including malignant thymoma, or myeloproliferative or lymphoproliferative disorders at any time, unless deemed cured by adequate treatment with no evidence of recurrence for ≥5 years before Screening. Patients with completely excised nonmelanoma skin cancers (such as basal cell carcinoma or squamous cell carcinoma) or cervical carcinoma in situ would be permitted at any time.
12. Have a history of cerebrovascular accident or myocardial infarction within the last 12 months before Screening, or current severe/unstable angina, arrhythmia, symptomatic congestive heart failure New York Heart Association (NYHA) class III or IV, or uncontrolled hypertension.
13. Have clinical evidence of significant unstable or uncontrolled acute or chronic diseases (i.e., cardiovascular, pulmonary, hematologic, gastrointestinal, endocrinologic, hepatic, renal, neurologic, malignancy, or infectious diseases) which, in the opinion of the Investigator, could confound the results of the study or put the patient at undue risk.
14. Major past surgery (e.g., heart valve replacement, hip replacement) that, in the opinion of the Investigator, poses a risk to patient's safety or interferes with the study evaluation, procedures or completion.
15. Thymectomy when performed < 3 months prior to Screening.
16. History or presence of alcoholism or drug/chemical/substance abuse within 2 years before Screening per Investigator's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-12-30 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2017-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Guglietta, MD, Study Director — argenx
Locations (19):
- United States (6):
  - Investigator Site 19, Irvine, California
  - Investigator Site 17, Los Angeles, California
  - Investigator Site 15, Tampa, Florida
  - Investigator Site 16, Indianapolis, Indiana
  - Investigator Site 14, Chapel Hill, North Carolina
  - Investigator Site 18, Dublin, Ohio
- Belgium (2):
  - Investigator Site 2, Ghent
  - Investigator Site 1, Leuven
- Canada (2):
  - Investigator Site 4, Montreal
  - Investigator Site 3, Toronto
- Italy (3):
  - Investigator Site 7, Bergamo
  - Investigator Site 6, Milan
  - Investigator Site 5, Roma
- Investigator Site 8, Leiden, Netherlands
- Poland (2):
  - Investigator Site 10, Gdansk
  - Investigator Site 9, Krakow
- Spain (2):
  - Investigator Site 12, Barcelona
  - Investigator Site 11, Madrid
- Investigator Site 13, Solna, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 30 December 2016, 15 study centers in 8 countries (Belgium, Canada, Italy, the Netherlands, Poland, Spain, Sweden, and United States) consented at least 1 patient with myasthenia gravis (MG) who had generalized muscle weakness. The last patient last visit was 20 October 2017.
Pre-assignment Details: The study included a maximum screening period of 15 days to evaluate patients' eligibility. Eligible patients were randomized in a 1:1 ratio to receive either ARGX-113 at 10 milligram/ kilogram (mg/kg) body weight or placebo, in addition to Standard of Care (SoC). The study involved a 3-week treatment period and an 8-week follow-up period.
Groups:
- ARGX-113: Patients received ARGX-113 at a dose of 10 mg/kg in 4 intravenous (IV) infusions, administered 1 week apart, in addition to SoC.
- Placebo: Patients received matching placebo in 4 IV infusions, administered 1 week apart, in addition to SoC.
Period: Overall Study
Arm/Group | ARGX-113 | Placebo
Started | 12 | 12
Completed | 11 | 12
Not Completed | 1 | 0
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are summarized for the randomized population which included patients who had been allocated to a randomized treatment group, regardless of whether they received the planned treatment or not.
Groups:
- ARGX-113: Patients received ARGX-113 at a dose of 10 mg/kg in 4 IV infusions, administered 1 week apart, in addition to SoC.
- Total: Total of all reporting groups
Arm/Group | ARGX-113 | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 10 | 18
  >=65 years | 4 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (13.60) | 43.5 (19.28) | 49.4 (17.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 12 | 23
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 11 | 11 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Weight [Mean (Standard Deviation); unit: kg] | 74.08 (15.477) | 75.21 (14.343) | 74.64 (14.604)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment Emergent Adverse Events (TEAES) and Treatment Emergent Serious Adverse Events (SAEs)
Description: TEAEs were defined as AEs that first occurred or worsened in severity after the first administration of the treatment. A treatment emergent SAE was any untoward medical occurrence that resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization;resulted in persistent or significant disability or incapacity; was a congenital abnormality or birth defect; or other medically significant events. All TEAEs observed were graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03 with descriptions of severity for each AE based on the following general guideline: Grade 1= mild; Grade 2 = moderate; Grade 3 = severe or medically significant but not immediately life-threatening; Grade 4 = life-threatening consequences; Grade 5 = death related to AE.
Time Frame: Day 1 to Day 78
Population: The safety analysis set included all patients in the randomized population who received at least 1 dose or part of a dose. The safety analysis was based on the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | ARGX-113 | Placebo
Number analyzed (Participants) | 12 | 12
Participants
  At least 1 TEAE | 10 | 10
  At least 1 treatment-related TEAE | 8 | 3
  At least 1 treatment emergent SAE | 0 | 0
  Withdrawn from treatment with at least 1 TEAE | 0 | 0
  Discontinued study due to at least 1 TEAE | 0 | 0
  NCI-CTCAE severity Grade ≥3 | 0 | 0
  Number of Deaths | 0 | 0

2. Primary Outcome: Mean Change From Baseline in Vital Signs: Blood Pressure
Description: The patients' diastolic and systolic blood pressure were measured pre-dose on dosing days 1,8,15 and 22 and also during the follow up period. The mean change from baseline at each time point is presented. Baseline is defined as the last non-missing value before first dose of study medication.
Time Frame: Baseline and Days 8,15, 22, 29, 36, 43, 50, 64 and 78
Population: The safety analysis set included all patients in the randomized population who received at least 1 dose or part of a dose. The safety analysis was based on the actual treatment received.
  Only patients with data available for analysis are presented.
Measure: Mean (Standard Deviation); unit: millimeters mercury
Arm/Group | ARGX-113 | Placebo
Number analyzed (Participants) | 12 | 12
millimeters mercury
  Systolic- Day 8 | 3.8 (9.12) | 6.3 (10.52)
  Systolic- Day 15 | 4.5 (15.62) | 2.7 (10.97)
  Systolic- Day 22 | 2.7 (9.30) | 3.0 (13.03)
  Systolic- Day 29: number analyzed (Participants) | 12 | 11
  Systolic- Day 29 | 8.2 (10.70) | 1.2 (9.06)
  Systolic- Day 36 | 8.5 (12.93) | 3.2 (5.41)
  Systolic- Day 43: number analyzed (Participants) | 12 | 11
  Systolic- Day 43 | 5.4 (12.47) | 4.6 (8.27)
  Systolic- Day 50: number analyzed (Participants) | 11 | 10
  Systolic- Day 50 | 10.6 (9.78) | 6.6 (12.58)
  Systolic- Day 64: number analyzed (Participants) | 10 | 12
  Systolic- Day 64 | 4.3 (10.41) | 0.1 (14.84)
  Systolic- Day 78: number analyzed (Participants) | 11 | 12
  Systolic- Day 78 | 2.5 (10.82) | 6.8 (10.33)
  Diastolic- Day 8 | -0.8 (7.48) | -0.3 (10.55)
  Diastolic- Day 15 | 1.5 (9.58) | -0.8 (9.34)
  Diastolic- Day 22 | -0.3 (6.01) | -2.3 (10.52)
  Diastolic- Day 29: number analyzed (Participants) | 12 | 11
  Diastolic- Day 29 | 4.0 (8.95) | -4.4 (11.89)
  Diastolic- Day 36 | 3.6 (11.73) | -0.3 (6.80)
  Diastolic- Day 43: number analyzed (Participants) | 12 | 11
  Diastolic- Day 43 | 2.9 (6.95) | -5.1 (10.09)
  Diastolic- Day 50: number analyzed (Participants) | 11 | 10
  Diastolic- Day 50 | 4.7 (7.38) | -0.5 (16.39)
  Diastolic- Day 64: number analyzed (Participants) | 10 | 12
  Diastolic- Day 64 | 3.1 (4.77) | -4.7 (8.96)
  Diastolic- Day 78: number analyzed (Participants) | 11 | 12
  Diastolic- Day 78 | 1.7 (7.28) | -3.5 (10.41)

3. Primary Outcome: Mean Change From Baseline in Vital Signs: Heart Rate
Description: The patients' heart rate was measured pre-dose on dosing days 1,8,15 and 22 and also during the follow up period. The mean change from baseline at each time point is presented. Baseline is defined as the last non-missing value before first dose of study medication.
Time Frame: Baseline and Days 8,15, 22, 29, 36, 43, 50, 64 and 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | ARGX-113 | Placebo
Number analyzed (Participants) | 12 | 12
beats/minute
  Day 8 | -2.7 (11.80) | 1.8 (11.66)
  Day 15 | -4.1 (9.05) | 2.5 (12.40)
  Day 22 | -0.8 (10.70) | -1.1 (12.15)
  Day 29: number analyzed (Participants) | 12 | 11
  Day 29 | -2.4 (13.49) | 0.1 (9.75)
  Day 36 | 1.1 (14.08) | 3.1 (11.87)
  Day 43: number analyzed (Participants) | 12 | 11
  Day 43 | 0.2 (10.79) | 3.1 (15.49)
  Day 50: number analyzed (Participants) | 11 | 10
  Day 50 | 0.5 (19.82) | 2.1 (12.98)
  Day 64: number analyzed (Participants) | 10 | 12
  Day 64 | -4.0 (19.22) | 0.6 (8.71)
  Day 78: number analyzed (Participants) | 11 | 12
  Day 78 | -3.1 (10.78) | -2.0 (15.12)

4. Primary Outcome: Mean Change From Baseline in Vital Signs: Temperature
Description: The patients' temperature was measured pre-dose on dosing days 1,8,15 and 22 and also during the follow up period. The mean change from baseline at each time point is presented. Baseline is defined as the last non-missing value before first dose of study medication.
Time Frame: Baseline and Days 8,15, 22, 29, 36, 43, 50, 64 and 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees Centigrade
Arm/Group | ARGX-113 | Placebo
Number analyzed (Participants) | 12 | 12
degrees Centigrade
  Day 8 | 0.18 (0.493) | 0.15 (0.511)
  Day 15 | 0.09 (0.535) | 0.16 (0.382)
  Day 22 | 0.05 (0.613) | 0.27 (0.429)
  Day 29: number analyzed (Participants) | 12 | 11
  Day 29 | -0.03 (0.459) | 0.11 (0.291)
  Day 36 | -0.13 (0.620) | 0.09 (0.334)
  Day 43: number analyzed (Participants) | 12 | 11
  Day 43 | -0.04 (0.563) | 0.08 (0.299)
  Day 50: number analyzed (Participants) | 11 | 10
  Day 50 | -0.03 (0.341) | 0.10 (0.422)
  Day 64: number analyzed (Participants) | 9 | 12
  Day 64 | 0.21 (0.593) | 0.17 (0.306)
  Day 78: number analyzed (Participants) | 11 | 12
  Day 78 | 0.11 (0.552) | 0.18 (0.282)

5. Primary Outcome: Mean Change From Baseline in Vital Signs: Weight
Description: The patients' weight as measured pre-dose on dosing days 1,8,15 and 22 and also during the follow up period. The mean change from baseline at each time point is presented. Baseline is defined as the last non-missing value before first dose of study medication.
Time Frame: Baseline and Days 8,15, 22, 29, 36, 43, 50, 64 and 78
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | ARGX-113 | Placebo
Number analyzed (Participants) | 12 | 12
kg
  Day 8 | 0.18 (0.443) | -0.02 (1.359)
  Day 15 | 0.60 (0.768) | 0.31 (1.528)
  Day 22 | 0.54 (0.672) | 0.01 (1.672)
  Day 29: number analyzed (Participants) | 12 | 11
  Day 29 | 0.41 (0.729) | -0.04 (1.826)
  Day 36 | 0.76 (0.840) | -0.02 (1.770)
  Day 43: number analyzed (Participants) | 12 | 11
  Day 43 | 0.91 (2.093) | 0.31 (2.593)
  Day 50: number analyzed (Participants) | 11 | 9
  Day 50 | 0.48 (1.156) | 0.44 (1.996)
  Day 64: number analyzed (Participants) | 10 | 12
  Day 64 | 0.26 (1.052) | -0.27 (2.703)
  Day 78: number analyzed (Participants) | 11 | 12
  Day 78 | 0.23 (1.238) | -0.60 (3.122)

6. Primary Outcome: Number of Patients With Abnormal Clinically Relevant Findings in Electrocardiogram (ECG) Parameters
Description: ECG parameters of heart rate, PR, QT, and QRS interval were read locally and performed pre-dose on dosing days 1,8,15 and 22 and on the last follow up visit on Day 78. Any patients recording abnormal clinically relevant findings during the study are presented.
Time Frame: Day 1 to Day 78
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ARGX-113 | Placebo
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

7. Primary Outcome: Number of Patients With Abnormal Clinical Laboratory Findings Reported as TEAEs
Description: Sampling for clinical laboratory tests including hematology, clinical chemistry, and urinalysiswas performed pre-dose on dosing Days 1, 8, 15 and 22 and throughout the follow up period. Patients fasted for at least 8 hours prior to this sampling. Abnormal laboratory values, or test results were not reported as TEAEs unless they were associated with clinical signs and symptoms that were considered clinically relevant, required therapy or led to treatment discontinuation. Patients reporting TEAEs in any of the laboratory parameters during the study are presented.
Time Frame: Day 1 to Day 78
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ARGX-113 | Placebo
Number analyzed (Participants) | 12 | 12
Participants
  B-lymphocyte count decreased | 2 | 0
  T-lymphocyte count decreased | 1 | 0
  Lymphocyte count decreased | 2 | 0
  Monocyte count decreased | 2 | 0
  Neutrophil count inceased | 2 | 0
  Blood thyroid stimulating hormone increased | 1 | 0

8. Secondary Outcome: Mean Change From Baseline in Myasthenia Gravis-Activities of Daily Living (MG-ADL) Score
Description: The MG-ADL is an 8-item patient-reported scale to assess MG symptoms and their effects on daily activities. It evaluates the capacity to perform different activities of daily living such as talking, chewing, swallowing, breathing, brushing the teeth/combing the hair, or arising from the chair and it also assesses double vision and eyelid droop. The 8 items are rated from 0 to 3 and the total score could point from 0 to 24; with higher scores indicating more impairment. The mean change in MG-ADL score from baseline is presented for each timepoint with a clinically meaningful improvement defined as a drop of at least 2 points as compared with baseline.
Time Frame: Baseline and Days 8,15, 22, 29, 36, 43, 50, 64 and 78
Population: The full analysis set (FAS) included all randomized patients with at least 1 of the MG-ADL, Quantitative Myasthenia Gravis (QMG), Myasthenia Gravis Composite (MGC), and 15-item Quality of Life scale for Myasthenia Gravis revised version (MGQoL15r) scales available for 1 of the postbaseline assessments up to Day 78 along with the corresponding baseline value. Only patients with data available for analysis are presented.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARGX-113 | Placebo
Number analyzed (Participants) | 12 | 12
score on a scale
  Day 8 | -1.9 (2.75) | -0.7 (1.56)
  Day 15 | -2.8 (2.70) | -2.2 (2.08)
  Day 22 | -3.5 (2.84) | -2.5 (2.50)
  Day 29: number analyzed (Participants) | 12 | 11
  Day 29 | -4.1 (2.64) | -2.3 (2.72)
  Day 36 | -4.2 (3.30) | -2.1 (2.43)
  Day 43: number analyzed (Participants) | 12 | 11
  Day 43 | -3.8 (2.72) | -2.4 (2.69)
  Day 50: number analyzed (Participants) | 11 | 10
  Day 50 | -4.4 (3.53) | -2.9 (2.96)
  Day 64: number analyzed (Participants) | 10 | 12
  Day 64 | -3.4 (3.27) | -1.8 (3.55)
  Day 78: number analyzed (Participants) | 11 | 12
  Day 78 | -3.5 (3.50) | -1.8 (4.22)

9. Secondary Outcome: Mean Change From Baseline in QMG Score
Description: The QMG quantifies disease severity based on impairments of body functions and structures as defined by the International Classification of Disability and Health.
  The QMG consists of 13 items that includes ocular, bulbar, and limb function. Out of the 13 items, 6 are timed tests of endurance measured in seconds. Each item has a possible score from 0-3. The score range is 0-39, where higher scores indicate more severe impairments. The mean change in QMG score from baseline is presented with a clinically meaningful improvement defined as a drop of at least 3 points as compared with baseline.
Time Frame: Baseline and Days 8,15, 22, 29, 36, 43, 50, 64 and 78
Population: The FAS includes all randomized patients with at least 1 of the MG-ADL, QMG, MGC, and MGQoL15r scales available for 1 of the postbaseline assessments up to Day 78 along with the corresponding baseline value. Only patients with data available for analysis are presented.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARGX-113 | Placebo
Number analyzed (Participants) | 12 | 12
score on a scale
  Day 8 | -2.8 (3.13) | 0.0 (2.22)
  Day 15 | -4.0 (4.29) | -1.8 (3.08)
  Day 22 | -4.0 (4.55) | -1.8 (3.91)
  Day 29: number analyzed (Participants) | 12 | 11
  Day 29 | -4.9 (4.94) | -1.4 (3.72)
  Day 36 | -5.7 (5.97) | -1.9 (3.37)
  Day 43: number analyzed (Participants) | 12 | 11
  Day 43 | -4.6 (5.73) | -2.1 (4.55)
  Day 50: number analyzed (Participants) | 10 | 9
  Day 50 | -5.5 (5.84) | -2.1 (3.95)
  Day 64: number analyzed (Participants) | 10 | 10
  Day 64 | -4.5 (6.42) | -1.8 (4.59)
  Day 78: number analyzed (Participants) | 10 | 10
  Day 78 | -4.8 (7.67) | -2.1 (5.07)

10. Secondary Outcome: Mean Change From Baseline in MGC Score
Description: The MGC has 10 items combining physician examination and patient-reported outcomes. The 2 ocular items are derived from QMG. It has 3 items on muscle strength (deltoids, hip flexors, and neck flexors or extensors) and 4 items on bulbar function (swallowing, chewing, breathing, and speech functions), based on the clinical history. Each item is scored on an ordinal scale with 4 possible categories, but the items are weighted, whereby bulbar impairments weigh more than ocular ones. The impairments that were examined by the Investigator included ptosis or upward gaze, double vision, eye closure, neck flexion, shoulder abduction, and hip flexion. The patient-reported outcomes under MGC are talking, chewing, swallowing, and breathing. The maximum possible score is 50 (range from 0-50), with higher scores reflecting more severe impairments. The mean change in MGC score from baseline is presented.
Time Frame: Baseline and Days 8,15, 22, 29, 36, 43, 50, 64 and 78
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARGX-113 | Placebo
Number analyzed (Participants) | 12 | 12
score on a scale
  Day 8 | -4.3 (5.87) | -1.3 (2.77)
  Day 15 | -5.8 (6.45) | -4.4 (4.56)
  Day 22 | -7.8 (6.92) | -4.0 (3.86)
  Day 29: number analyzed (Participants) | 12 | 11
  Day 29 | -8.7 (7.36) | -4.1 (5.22)
  Day 36 | -9.0 (8.73) | -4.1 (5.58)
  Day 43: number analyzed (Participants) | 12 | 11
  Day 43 | -8.6 (8.54) | -3.5 (5.97)
  Day 50: number analyzed (Participants) | 11 | 10
  Day 50 | -9.4 (7.92) | -4.2 (5.51)
  Day 64: number analyzed (Participants) | 10 | 12
  Day 64 | -7.2 (8.65) | -3.8 (6.84)
  Day 78: number analyzed (Participants) | 11 | 12
  Day 78 | -7.1 (9.71) | -3.8 (6.83)

11. Secondary Outcome: Mean Change From Baseline in MGQoL15r Score
Description: The MGQoL15r is a quality of life scale or survey of patient's responses that addresses MG-specific psychological well-being and social functioning. It is a brief questionnaire that is completed by the patient and uses 3 response options to help inform the clinician about the patient's perception of the extent of and dissatisfaction with MG-related dysfunction. Each item is scored from 0 to 2 according to its frequency, with a maximum score of 30 (range 0-30) and higher scores reflecting more severe impairment. The mean change in MGQoL15r score from baseline is presented.
Time Frame: Baseline and Days 8,15, 22, 29, 36, 43, 50, 64 and 78
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARGX-113 | Placebo
Number analyzed (Participants) | 12 | 12
score on a scale
  Day 8 | -2.0 (5.77) | -0.8 (1.86)
  Day 15 | -3.7 (4.42) | -1.0 (2.76)
  Day 22: number analyzed (Participants) | 12 | 11
  Day 22 | -4.3 (4.77) | -1.5 (3.17)
  Day 29: number analyzed (Participants) | 11 | 11
  Day 29 | -4.7 (5.44) | -1.5 (2.91)
  Day 36: number analyzed (Participants) | 11 | 12
  Day 36 | -6.0 (5.78) | -2.1 (3.58)
  Day 43: number analyzed (Participants) | 12 | 11
  Day 43 | -5.3 (5.59) | -1.4 (3.70)
  Day 50: number analyzed (Participants) | 11 | 10
  Day 50 | -4.4 (4.13) | -1.8 (3.71)
  Day 64: number analyzed (Participants) | 10 | 12
  Day 64 | -3.7 (5.10) | -1.3 (3.68)
  Day 78: number analyzed (Participants) | 11 | 12
  Day 78 | -2.7 (5.44) | -1.5 (3.61)

12. Secondary Outcome: Maximum Reduction From Baseline in MG-ADL Score
Description: The MG-ADL is an 8-item patient-reported scale to assess MG symptoms and their effects on daily activities. It evaluates the capacity to perform different activities of daily living such as talking, chewing, swallowing, breathing, brushing the teeth/combing the hair, or arising from the chair and it also assesses double vision and eyelid droop. The 8 items are rated from 0 to 3 and the total score could point from 0 to 24; with higher scores indicating more impairment. The mean maximum reduction from baseline across all visit days for MG-ADL score is presented.
Time Frame: Day 1 to Day 78
Population: The FAS includes all randomized patients with at least 1 of the MG-ADL, QMG, MGC, and MGQoL15r scales available for 1 of the postbaseline assessments up to Day 78 along with the corresponding baseline value.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARGX-113 | Placebo
Number analyzed (Participants) | 12 | 12
score on a scale | -5.1 (3.32) | -3.7 (2.93)

13. Secondary Outcome: Maximum Reduction From Baseline in QMG Score
Description: The QMG quantifies disease severity based on impairments of body functions and structures as defined by the International Classification of Disability and Health.
  The QMG consists of 13 items that included ocular, bulbar, and limb function. Out of the 13 items, 6 are timed tests of endurance measured in seconds. Each item has a possible score from 0-3. The total possible score is 39 (range 0-39), where higher scores indicates more severe impairments. The mean maximum reduction from baseline across all visit days for QMG score is presented.
Time Frame: Day 1 to Day 78
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARGX-113 | Placebo
Number analyzed (Participants) | 12 | 12
score on a scale | -7.3 (6.08) | -4.3 (4.16)

14. Secondary Outcome: Maximum Reduction From Baseline in MGC Score
Description: The MGC has 10 items combining physician examination and patient-reported outcomes. The 2 ocular items are derived from QMG. It has 3 items on muscle strength (deltoids, hip flexors, and neck flexors or extensors) and 4 items on bulbar function (swallowing, chewing, breathing, and speech functions), based on the clinical history. Each item is scored on an ordinal scale with 4 possible categories, but the items are weighted, whereby bulbar impairments weigh more than ocular ones. The impairments that were examined by the Investigator included ptosis or upward gaze, double vision, eye closure, neck flexion, shoulder abduction, and hip flexion. The patient-reported outcomes under MGC are talking, chewing, swallowing, and breathing. The maximum possible score is 50 (range 0-50), with higher scores reflecting more severe impairments. The mean maximum reduction from baseline across all visit days for MCG score is presented.
Time Frame: Day 1 to Day 78
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARGX-113 | Placebo
Number analyzed (Participants) | 12 | 12
score on a scale | -11.5 (7.61) | -7.7 (4.40)

15. Secondary Outcome: Maximum Reduction From Baseline in MGQoL15r Score
Description: The MGQoL15r is a quality of life scale or survey of patient's responses that addresses MG-specific psychological well-being and social functioning. It is a brief questionnaire that was completed by the patient and uses 3 response options to help inform the clinician about the patient's perception of the extent of and dissatisfaction with MG-related dysfunction. Each item is scored from 0 to 2 according to its frequency, with a maximum score of 30 (range 0-30) and higher scores reflecting more severe impairment. The mean maximum reduction from baseline across all visit days for MGQoL15r score is presented.
Time Frame: Day 1 to Day 78
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ARGX-113 | Placebo
Number analyzed (Participants) | 12 | 12
score on a scale | -7.2 (5.42) | -3.0 (3.16)

16. Secondary Outcome: Pharmacokinetic (PK) Parameters - Plasma Concentrations of ARGX-113
Description: The appropriate PK parameters were calculated after single (Day 1) and multiple administrations (Days 8,15 and 22) of ARGX-113. The mean maximum observed plasma concentration (Cmax) and plasma concentration observed pre-dose (Ctrough) is presented.
Time Frame: Days 1, 8, 15 and 22
Population: The PK analysis set included all patients in the randomized population who had at least 1 plasma concentration data value available for ARGX-113 without major protocol deviations thought to impact PK. Patients who did not receive ARGX-113 were not included in the PK analysis set. Only patients with data available for analysis are presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | ARGX-113
Number analyzed (Participants) | 12
nanograms/milliliter (ng/mL)
  Cmax - Day 1 | 179063.7 (31.9)
  Cmax - Day 8: number analyzed (Participants) | 11
  Cmax - Day 8 | 173960.4 (19.5)
  Cmax - Day 15: number analyzed (Participants) | 11
  Cmax - Day 15 | 153257.2 (22.1)
  Cmax - Day 22: number analyzed (Participants) | 11
  Cmax - Day 22 | 162655.6 (26.1)
  Ctrough - Day 1 | 7266.2 (43.5)
  Ctrough - Day 8: number analyzed (Participants) | 11
  Ctrough - Day 8 | 9894.8 (54.7)
  Ctrough - Day 15: number analyzed (Participants) | 11
  Ctrough - Day 15 | 10045.5 (56.7)
  Ctrough - Day 22: number analyzed (Participants) | 11
  Ctrough - Day 22 | 10944.6 (71.1)

17. Secondary Outcome: PK Parameters - Median Time of Occurrence of Cmax (Tmax) of ARGX-113
Description: The appropriate PK parameters were calculated after single (Day 1) and multiple administrations (Days 8, 15 and 22) of ARGX-113. The median tmax is presented.
Time Frame: Days 1, 8 15 and 22.
Population: as for outcome 16
Measure: Median (Full Range); unit: hours
Arm/Group | ARGX-113
Number analyzed (Participants) | 12
hours
  Day 1 | 2.44 [2.08 to 2.58]
  Day 8 | 2.50 [2.08 to 2.50]
  Day 15 | 2.50 [2.07 to 2.50]
  Day 22 | 2.46 [2.08 to 2.67]

18. Secondary Outcome: PK Parameters - Apparent Terminal Half-life (t1/2 Lambda z) of ARGX-113
Description: The t1/2 lambda z was calculated at Day 22.
Time Frame: Day 22
Population: The PK analysis set included all patients in the randomized population who had at least 1 plasma concentration data value available for ARGX-113 without major protocol deviations thought to impact PK. Patients who did not receive ARGX-113 were not included in the PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | ARGX-113
Number analyzed (Participants) | 12
hours | 116.08 (15.8)

19. Secondary Outcome: PK Parameters - Accumulation Ratio (Rac) of ARGX-113
Description: The Rac was calculated as Day 22 Cmax/Day 1 Cmax.
Time Frame: Days 1 and 22.
Population: The PK analysis set included all patients in the randomized population who had at least 1 plasma concentration data value available for ARGX-113 without major protocol deviations thought to impact PK. Patients who did not receive ARGX-113 were not included in the PK analysis set. Only patinents with data available for analysis are presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | ARGX-113
Number analyzed (Participants) | 11
ratio | 0.9360 (25.7)

20. Secondary Outcome: Mean Percent Change From Baseline in Immunoglobulins (IgGs)
Description: The pharmacodynamic (PD) biomarkers that were measured included the following IgGs: Total IgG and IgG isotypes; IgG1, IgG2, IgG3, IgG4. PD samples were collected pre-dose on dosing days and the mean percent change from baseline at the end of treatment (Day 22) and at the last follow up visit (Day 78) are presented.
Time Frame: Baseline, Days 22 and 78
Population: The PD analysis set included all patients in the randomized population who had at least 1 non-missing post-dose PD measurement available without major protocol deviations thought to impact PD. Only patients with data available for analysis are presented.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | ARGX-113 | Placebo
Number analyzed (Participants) | 12 | 12
percentage change
  Total IgG - Day 22 | -70.0 (10.96) | -2.8 (15.34)
  Total IgG - Day 78 | -20.4 (24.96) | 6.4 (27.49)
  IgG1 - Day 22 | -65.5 (8.56) | -2.1 (9.29)
  IgG1 - Day 78 | -16.0 (18.17) | -1.1 (19.01)
  IgG2 - Day 22 | -61.0 (6.73) | -4.4 (6.99)
  IgG2 - Day 78 | -34.9 (16.02) | -5.3 (17.63)
  IgG3 - Day 22 | -65.25 (10.045) | 0.57 (9.566)
  IgG3 - Day 78 | -5.19 (18.422) | 2.52 (15.341)
  IgG4 - Day 22 | -49.48 (10.278) | 0.79 (6.592)
  IgG4 - Day 78 | 4.16 (25.513) | 1.57 (16.730)

21. Secondary Outcome: Mean Percent Change From Baseline in Anti-Acetylcholine Receptor (AChR) Antibodies
Description: Analysis of the PD biomarkers included anti-AChR binding antibodies. PD samples were collected pre-dose on dosing days and the mean percent change from baseline at the end of treatment (Day 22) and at the last follow up visit (Day 78) are presented.
Time Frame: Baseline, Days 22 and 78
Population: The PD analysis set includes all patients in the randomized population who had at least 1 non-missing post-dose PD measurement available without major protocol deviations thought to impact PD. Only patients with data available for analysis are presented.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | ARGX-113 | Placebo
Number analyzed (Participants) | 12 | 12
percentage change
  Day 22 | -52.2686 (26.32992) | -0.3236 (8.50886)
  Day 78 | -1.3361 (34.33867) | -7.8881 (33.43325)

22. Secondary Outcome: Number of Patients With an Anti-drug Antibodies (ADA) Response
Description: Blood samples to assess ADA were collected pre-dose on dosing days and throughout the follow up period. The overall number of patients with pre-dose and post-dose ADA titers are presented.
Time Frame: Baseline up to Day 78
Population: The PD analysis set included all patients in the randomized population who had at least 1 non-missing post-dose PD measurement available without major protocol deviations thought to impact PD.
Measure: Number; unit: participants
Arm/Group | ARGX-113 | Placebo
Number analyzed (Participants) | 12 | 12
participants
  Patients with pre-dose ADA titers | 4 | 2
  Patients with post-dose ADA titers | 4 | 3

ADVERSE EVENTS:
Time Frame: Day 1 to Day 78.
Description: TEAEs were monitored continuously from Day 1 until last study-related activity. In case of early discontinuation, any TEAEs were assessed for 30 days following the patient's last visit or until satisfactory resolution or stabilization. The safety analysis set included patients in the randomized population who received at least 1 dose or part of a dose. The safety analysis was based on the actual treatment received.
Arm/Group | ARGX-113 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 10/12 | 10/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARGX-113 (N=12) | Placebo (N=12)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (9) | 3 (5)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 2 (3)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (2)
Infusion site pain (General disorders) | 1 (1) | 0 (0)
Infusion site pruritus (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
B-lymphocyte count decreased (Investigations) | 2 (3) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (4) | 0 (0)
Monocyte count decreased (Investigations) | 2 (4) | 0 (0)
Neutrophil count increased (Investigations) | 2 (4) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0)
T-lymphocyte count decreased (Investigations) | 1 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Premenstrual headache (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-11-28): https://cdn.clinicaltrials.gov/large-docs/73/NCT02965573/Prot_002.pdf
  • Statistical Analysis Plan (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT02965573/SAP_001.pdf